CLINICAL TRIAL: NCT02981641
Title: Intraoperative Radiotherapy (IORT) Versus Concurrent Chemoradiotherapy (CCRT) for Pancreatic Cancer
Brief Title: IORT Versus CCRT for Pancreatic Cancer
Acronym: IVCPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Chengfeng Wang, Director of Department of Abdominal Surgical Oncolgoy, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012AA022701
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-11

CONDITIONS: Pancreatic Cancer Stage IV
Keywords: Pancreatic cancer; Intraoperative radiotherapy (IORT); Concurrent Chemoradiotherapy (CCRT)
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiotherapy, Conformal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intraoperative radiotherapy (IORT) Group (Experimental): Radiotherapy (Total dose: 18~22 Gy; Single dose: 18~22 Gy; Frequency: 1) + Sequential chemotherapy
  Interventions: Radiation: Intraoperative radiotherapy (IORT); Drug: Sequential chemotherapy
- Concurrent Chemoradiotherapy (CCRT) Group (Experimental): Three dimensional conformal radiation therapy (3D-CRT) (Total dose: 60 Gy; Single dose: 2 Gy; Frequency: 30) + Concurrent chemotherapy (Gemcitabine(GEM), 800 mg/m2 weekly on Day 1-21, Q28d; or S-1 orally, 400 mg/d, bid on Day 1-21, Q28d) + Sequential chemotherapy
  Interventions: Drug: Sequential chemotherapy; Radiation: Three dimensional conformal radiation therapy (3D-CRT); Drug: Concurrent chemotherapy

INTERVENTIONS:
Radiation: Intraoperative radiotherapy (IORT) — Total dose: 18~22 Gy; Single dose: 18~22 Gy; Frequency: 1
  Other Names: IORT
  Arms: Intraoperative radiotherapy (IORT) Group
Drug: Sequential chemotherapy — Sequential chemotherapy
  Other Names: SC
Radiation: Three dimensional conformal radiation therapy (3D-CRT) — Total dose: 60 Gy; Single dose: 2 Gy; Frequency: 30
  Other Names: 3D-CRT
  Arms: Concurrent Chemoradiotherapy (CCRT) Group
Drug: Concurrent chemotherapy — Gemcitabine (GEM), 800 mg/m2 weekly on Day 1-21, Q28d; or S-1 orally, 400 mg/d, bid on Day 1-21, Q28d
  Other Names: CC
  Arms: Concurrent Chemoradiotherapy (CCRT) Group

SUMMARY:
The purpose of this study is to find the better radiation therapy between intraoperative radiotherapy (IORT) and concurrent chemoradiotherapy (CCRT).

DETAILED DESCRIPTION:
The trial is funded by National High-tech R&D Program (863 Program). The trial is prepared to be registered on the clinicaltrail.gov.

Quality assurance plan: Every participant is enrolled or excluded by two practiced investigators. And two investigators participated in all steps of the trail, including the record of the data, and the investigators will compare the data. If the data is consistent, the investigators would record the data; if not, the data would be checked and decided by the two investigators. All the steps and data are site monitored and audited by the workers of research and financial department of The First Affiliated Hospital of China Medical University Data check: The investigators compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry. Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources, including medical records and electronic case report forms. Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information, and normal ranges if relevant. Standard Operating Procedures to address registry operations and analysis activities, such as participants recruitment, data collection, data management, data analysis, reporting for adverse events, and change management. All registry operations would be done according to specific steps, and by two practiced investigators. Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect. According to the formula to differ advantages and disadvantages, the investigators need at least 100 participants to take part in the trail. The investigators can recruit about 120 participants every year according to previous experiences, so the investigators should recruit at least for one years.

Plan for missing data: The investigators would collect as much data as possible, and the investigators exclude the participants who cannot cooperate on recruitment. And the investigators manage situations according to statistical principles where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results.

Statistical analysis plan: Kaplan-Meier method would be used to analyze the difference of survival time between the two groups, and the local control rate of the two groups would be compared by chi square test. Statistical analyses would be performed by using IBM SPSS Statistics(version 20; IBM, Chicago, USA). The level of significance is defined as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as locally advanced pancreatic cancer.
* Cannot be treated by surgical resection.

Exclusion Criteria:

* Treated by chemotherapy or radiotherapy before.
* With distant organ metastasis.
* Cannot tolerate surgery (Intraoperative radiotherapy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Overal survival | 3 years
  OS

SECONDARY OUTCOMES:
Disease-specific survival | 3 years
  DSS
Progression-free survival | 3 years
  PFS
Local control rate | 3 years
  LCR

CONTACTS AND LOCATIONS:
Overall Officials: Chengfeng Wang, B.A., Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- CancerIHCAMS, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No